CLINICAL TRIAL: NCT03120481
Title: The Registry of Controls for Respiratory Diseases
Brief Title: Controls for Respiratory Diseases
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chang-Hoon Lee, Associate professor, Seoul National University Hospital
Other Study IDs: 2016-3435
Record Dates: First submitted 2017-04-14; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma; Idiopathic Pulmonary Fibrosis; Nontuberculous Mycobacterium Infection; Bronchiectasis; Lung Cancer
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Idiopathic Pulmonary Fibrosis; Mycobacterium Infections, Nontuberculous; Bronchiectasis; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — DNA Plasma Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normal control
  Interventions: Other: no intervation

INTERVENTIONS:
Other: no intervation — no intervention

SUMMARY:
This is the registry of control participants for patients with various respiratory diseases. We screened healthy volunteers who visited Seoul National Hospital Healthcare System Gangnam Center for routine health check-up, and enrolled patients who agree to participate in the study. The participants undergo baseline questionnaires, provide blood specimen and information of the results of health check-up. We will include participants as controls if they have no significant respiratory symptom and no significant radiographic abnormality. The data from this registry will be compared with those from other registry of various respiratory diseases

ELIGIBILITY:
Inclusion Criteria:

* 19-90 years old male and female
* underwent health check-up including chest radiography
* obtained informed consent

Exclusion Criteria:

* those who showed a significant abnormal finding of chest radiography
* those who reported a significant respiratory symptoms

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Those who visited the hospital for health check-up, and agree to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1572 (Estimated)
Dates: Start 2017-04-10 (Actual); Primary Completion 2037-02-28 (Estimated); Study Completion 2037-02-28 (Estimated)

PRIMARY OUTCOMES:
Mortality | 20 years
  Death

SECONDARY OUTCOMES:
Hospitalization | 20 years
  All cause hospitalization
Respiratory hospitalization | 20 years
  Hospitalization from respiratory causes
Respiratory diseases diagnosis | 20 years
  Respiratory diseases diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Hoon Lee, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Healthcare System Gangnam Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No